CLINICAL TRIAL: NCT00129246
Title: Naltrexone & Bupropion to Stop Smoking With Less Weight Gain
Brief Title: Low-Dose Naltrexone Combined With Bupropion to Stop Smoking With Less Weight Gain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAOMA15632-B; P50AA015632 (NIH); NIH Grant 9 P50-AA15632
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Smoking; Nicotine Dependence
Keywords: Tobacco; Smoking; Weight; Weight perception; Naltrexone; Bupropion
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Body Weight | interventions — Naltrexone; Bupropion

ARMS (2):
- Bupropion only (Active Comparator): The placebo comparator was a group of matched controls who received an identical psychosocial intervention and bupropion SR treatment regimen in a similar 7-week study investigation compared to naltrexone hydrochloride (25 mg/day) in combination with bupropion hydrochloride SR (300 mg/day).
  Interventions: Drug: Bupropion
- Naltrexone +Bupropion (Experimental): The active comparator in this 7-week open label study investigation was naltrexone hydrochloride (25 mg/day) in combination with bupropion hydrochloride SR (300 mg/day) compared to matched controls who received an identical psychosocial intervention and bupropion SR treatment regimen (bupropion only).
  Interventions: Drug: Naltrexone; Drug: Bupropion

INTERVENTIONS:
Drug: Naltrexone — Participants received naltrexone hydrochloride on the sixth day of bupropion treatment, and the initial dose was 12.5 mg, followed by 25 mg daily for the duration of the 7-week treatment.
  Arms: Naltrexone +Bupropion
Drug: Bupropion — Starting with the baseline visit, all participants received 150 mg of bupropion SR once per day for 3 days, then twice per day for the duration of the 7-week treatment period.

SUMMARY:
This study will test a combination of the drugs naltrexone and bupropion with weight-concerned smokers to investigate whether or not this combination of drugs improves smoking cessation quit rates and minimizes post quit weight gain.

DETAILED DESCRIPTION:
This is an open label smoking cessation clinical trial of 25 mg naltrexone with 300 mg bupropion sustained-release (SR) in six male and fourteen female participants. This pilot study is being conducted to determine:

* effect size estimates for smoking cessation and post-cessation weight gain, which will be used to compute the sample size needed for a large-scale clinical trial; and
* compliance with a combination of 25 mg naltrexone and 300 mg bupropion SR. In addition to examining the sample in this study, the investigators plan to compare this sample to a sample of matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Willingness and ability to give written consent
* Smoking at least 10 cigarettes per day for at least 1 year
* Baseline expired carbon-monoxide level of at least 10 ppm
* Weigh at least 100 lbs.
* English-speaking
* One person per household
* At least 1 prior quit attempt
* Concern about gaining weight. This will be assessed using a questionnaire that will provide a rating system to determine qualified participants.

Exclusion Criteria:

* Pregnant or nursing women or women attempting to conceive
* Serious current neurologic, psychiatric or medical illness, including unstable cardiac, hepatic, or renal disease and diabetes and hypertension
* Current alcohol dependence
* Current use of opiates, and/or a urine toxicology screen positive for opiates
* Chronic pain conditions necessitating opioid treatment (naltrexone, an opioid antagonist will make these medications ineffective)
* Evidence of significant hepatocellular injury as evidenced by AST or ALT >3 x normal or elevated bilirubin
* History of cirrhosis
* Body mass index (BMI) greater than 35
* History of anorexia nervosa or bulimia
* Current major depression
* Currently taking Toprol-XL (or metoprolol succinate)
* History of seizure disorder or serious brain injury
* Current use of smokeless tobacco, pipes, cigars, nicotine gum, nicotine patch, nicotine inhaler, nicotine lozenge, nicotine nasal spray, or bupropion
* Previous hypersensitivity to bupropion
* Patients requiring concomitant therapy with any psychotropic drug
* Participation in the Framing Messages for Smoking Cessation With Bupropion study (HIC#: 10880)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-12; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, Ph.D., Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Yale University School of Medicine Substance Abuse Treatment Unit, New Haven, Connecticut, United States

REFERENCES:
- [Result] Toll BA, Leary V, Wu R, Salovey P, Meandzija B, O'Malley SS. A preliminary investigation of naltrexone augmentation of bupropion to stop smoking with less weight gain. Addict Behav. 2008 Jan;33(1):173-9. doi: 10.1016/j.addbeh.2007.05.012. Epub 2007 Jun 2. PMID 17587504

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion Only: The placebo comparator was a group of matched controls who received an identical psychosocial intervention and bupropion SR treatment regimen in a similar 7-week study investigation compared to naltrexone hydrochloride (25 mg/day) in combination with bupropion hydrochloride SR (300 mg/day).
  Bupropion : Starting with the baseline visit, all participants received 150 mg of bupropion SR once per day for 3 days, then twice per day for the duration of the 7-week treatment period.
- Naltrexone +Bupropion: The active comparator in this 7-week open label study investigation was naltrexone hydrochloride (25 mg/day) in combination with bupropion hydrochloride SR (300 mg/day) compared to matched controls who received an identical psychosocial intervention and bupropion SR treatment regimen (bupropion only).
  Naltrexone : Participants received naltrexone hydrochloride on the sixth day of bupropion treatment, and the initial dose was 12.5 mg, followed by 25 mg daily for the duration of the 7-week treatment.
  Bupropion : Starting with the baseline visit, all participants received 150 mg of bupropion SR once per day for 3 days, then twice per day for the duration of the 7-week treatment period.
Period: Overall Study
Arm/Group | Bupropion Only | Naltrexone +Bupropion
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion Only | Naltrexone +Bupropion | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.3) | 43.0 (11.2) | 42.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation
Description: Smoking cessation is defined as the number of patients that displayed continuous 6-week abstinence from the quit date.
Time Frame: Week 6
Population: Per protocol analysis
Measure: Number; unit: participants
Arm/Group | Bupropion Only | Naltrexone +Bupropion
Number analyzed (Participants) | 20 | 20
participants | 6 | 6

2. Primary Outcome: Point Prevalence Abstinence
Description: Point prevalence abstinence is defined as the number of patients reporting point prevalence abstinence over the last 7 days.
Time Frame: Week 6
Population: Per protocol analysis
Measure: Number; unit: participants
Arm/Group | Bupropion Only | Naltrexone +Bupropion
Number analyzed (Participants) | 20 | 20
participants | 8 | 8

3. Secondary Outcome: Weight Gain Abstinent Participants
Description: Weight gain (in pounds) for the patients that were continuously abstinent at 6 weeks.
Time Frame: Week 6
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Bupropion Only | Naltrexone +Bupropion
Number analyzed (Participants) | 6 | 6
lbs | 3.17 (2.04) | 1.67 (3.17)

4. Primary Outcome: Weight Gain
Description: Weight gain for for the entire sample in pounds at 6 weeks.
Time Frame: Week 6
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Bupropion Only | Naltrexone +Bupropion
Number analyzed (Participants) | 20 | 20
lbs | 1.25 (2.90) | 0.28 (3.88)

ADVERSE EVENTS:
Arm/Group | Bupropion Only | Naltrexone +Bupropion
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion Only (N=20) | Naltrexone +Bupropion (N=20)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nervousness/anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 4 (4) | 4 (4)
Irritability (Psychiatric disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ringing in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No